CLINICAL TRIAL: NCT03261024
Title: Friction Versus Frictionless Mechanics During Maxillary En-masse Retraction in Adult Patients With Class I Bimaxillary Dentoalveolar Protrusion: A Randomized Clinical Trial
Brief Title: Friction Versus Frictionless Mechanics During Maxillary En-masse Retraction in Adult Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sally Magdi Riad, Assistant lecturer- Orthodontic department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Evidence based dentistry EBD
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: En-masse Retraction , Class I Bimaxillary Protrusion
Keywords: En-masse retraction , Class I bimaxillary protrusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Friction mechanics (Active Comparator): Upper and lower arches will be bonded, leveled and aligned until reaching 0.019 x 0.025 st st archwires.
  Miniscrews will be inserted in the buccal alveolar bone between second premolars and first molars bilaterally.
  Miniscrews will be connected to the molar bands by rigid wire. Extraction of upper first premolars. Upper anterior teeth will be ligated together. Hook between upper laterals and canines will be fixed on the main archwire.
  Nickel Titanium coil spring ( friction mechanics of retraction)will be used for maxillary en-masse retraction by extending the spring from the hook to the molar bands.
  Re-activation of the coil spring will be done in the follow up visits to maintain a constant force through the study.
  Interventions: Device: Friction mechanics
- Frictionless mechanics (Active Comparator): Upper and lower arches will be bonded, leveled and aligned until reaching 0.019 x 0.025 st st archwires.
  Miniscrews will be inserted in the buccal alveolar bone between second premolars and first molars bilaterally.
  Miniscrews will be connected to the molar bands by rigid wire. Extraction of upper first premolars. Upper anterior teeth will be ligated together. T-loops retraction arch ( frictionless mechanics of retraction)will be used for maxillary en-masse retraction. The wire will be cinched distal to the molar bands.
  Re-activation of the retraction loops will be done in the follow up visits to maintain a constant force through the study
  Interventions: Device: Frictionless mechanics

INTERVENTIONS:
Device: Friction mechanics — Nickel Titanium will be extended from the hook between the lateral incisors and canines to the first molar bands, to allow frictional en-masse retraction of anterior segment.
  Other Names: Nickel Titanium coil spring
  Arms: Friction mechanics
Device: Frictionless mechanics — T-loops retraction arch will be placed distal to the upper canines and cinched distal to the first molar bands, to allow frictionless en-masse retraction of anterior segment.
  Other Names: T-loops archwire
  Arms: Frictionless mechanics

SUMMARY:
This study is a Randomized clinical trial comparing the effectiveness of two different mechanics during maxillary en-masse retraction in adult patients. Patients will be randomly divided into two groups:Friction and frictionless mechanics. Mini screws will be used in both group to ensure maximum anchorage during retraction. Lateral cephalometric radiographs and dental models will be taken for each patients pre and post -retraction. Following complete anterior segment retraction, the rate and duration of retraction will be evaluated for both groups as well as patient satisfaction with treatment. Changes in incisors inclination and soft tissue as well as anchorage loss will be also assessed.

DETAILED DESCRIPTION:
Adult patients with Class I bimaxillary dentoalveolar protrusion will be recruited. All the patients need extraction of upper first premolars followed by anterior segment retraction and maximum anchorage.

The patients will be randomly allocated to one of two groups; either Friction or Frictionless group. In friction group, Nickel Titanium coil spring will be used for retraction of anterior segment while in frictionless group, T-loops will be used for retraction. All the patients will receive two miniscrews , one on each side to achieve maximum anchorage during retraction.

The patients will be seen on a monthly basis for follow up visit for activation of the appliance to maintain constant force during the study. An impression will be taken for the patients every visit, poured into stone for fabrication of dental models. The models will be used to monitor the rate of retraction of anterior teeth.

Every patient will be asked for lateral cephalometric radiograph before and after complete retraction. After data collection, two assessors will carry on the measurements blindly and independently. Statistical analysis of the data will be done and the results will be compared to evaluate the effectiveness of both techniques for en-masse retraction.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult patients with age range 18-30 yrs old.
2. Class I bimaxillary dentoalveolar protrusion .
3. Full permanent dentition.
4. Good oral hygiene.
5. Maximum anchorage is required.
6. Healthy bone between first molars and second premolars is needed.

Exclusion Criteria:

1. Systemic disease.
2. Severe crowding.
3. Extracted or missing upper permanent tooth/teeth (except for third molars).
4. Any signs or symptoms or previous history of temporomandibular disorders (TMD).
5. Previous orthodontic treatment.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Duration of retraction | After complete retraction, average 9 months
  months through clinical examination of the retracted anterior teeth
Rate of retraction | Average 9 months, recorded from the begin of retraction till the complete retraction of anterior teeth
  millimeters through dental models taken for each patient monthly at the follow up visit
Patient Satisfaction | After complete retraction , average 9 months
  Questionnaire will be filled by every patient at the end of the study regarding his experience and acceptance to the treatment, scale from 0 to 5 .

SECONDARY OUTCOMES:
Change in incisors inclination | After complete retraction, average 9 months
  Degree and millimeter through lateral cephalometric analysis
Change in soft tissue profile | After complete retraction, average 9 months
  Degree and millimeter through lateral cephalometric analysis
molar anchorage loss | After complete retraction, average 9 months
  Degree and millimeter through lateral cephalometric analysis

CONTACTS AND LOCATIONS:
Overall Officials: Fatma A. Abd El Sayed, Professor, Study Chair — Cairo University; Fady H. Fahim, lecturer, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
Participant information won't be used outside the study except with written permission of the participant

REFERENCES:
- [Background] Bills DA, Handelman CS, BeGole EA. Bimaxillary dentoalveolar protrusion: traits and orthodontic correction. Angle Orthod. 2005 May;75(3):333-9. doi: 10.1043/0003-3219(2005)75[333:BDPTAO]2.0.CO;2. PMID 15898369
- [Background] Park HS, Kwon TG. Sliding mechanics with microscrew implant anchorage. Angle Orthod. 2004 Oct;74(5):703-10. doi: 10.1043/0003-3219(2004)0742.0.CO;2. PMID 15529508
- [Background] Park HS, Yoon DY, Park CS, Jeoung SH. Treatment effects and anchorage potential of sliding mechanics with titanium screws compared with the Tweed-Merrifield technique. Am J Orthod Dentofacial Orthop. 2008 Apr;133(4):593-600. doi: 10.1016/j.ajodo.2006.02.041. PMID 18405824
- [Background] Upadhyay M, Yadav S, Patil S. Mini-implant anchorage for en-masse retraction of maxillary anterior teeth: a clinical cephalometric study. Am J Orthod Dentofacial Orthop. 2008 Dec;134(6):803-10. doi: 10.1016/j.ajodo.2006.10.025. PMID 19061808
- [Background] Heo W, Nahm DS, Baek SH. En masse retraction and two-step retraction of maxillary anterior teeth in adult Class I women. A comparison of anchorage loss. Angle Orthod. 2007 Nov;77(6):973-8. doi: 10.2319/111706-464.1. PMID 18004930
- [Background] Al-Sibaie S, Hajeer MY. Assessment of changes following en-masse retraction with mini-implants anchorage compared to two-step retraction with conventional anchorage in patients with class II division 1 malocclusion: a randomized controlled trial. Eur J Orthod. 2014 Jun;36(3):275-83. doi: 10.1093/ejo/cjt046. Epub 2013 Jun 20. PMID 23787192
- [Background] Felemban NH, Al-Sulaimani FF, Murshid ZA, Hassan AH. En masse retraction versus two-step retraction of anterior teeth in extraction treatment of bimaxillary protrusion. J Orthod Sci. 2013 Jan;2(1):28-37. doi: 10.4103/2278-0203.110330. PMID 24987640
- [Background] Ribeiro GL, Jacob HB. Understanding the basis of space closure in Orthodontics for a more efficient orthodontic treatment. Dental Press J Orthod. 2016 Mar-Apr;21(2):115-25. doi: 10.1590/2177-6709.21.2.115-125.sar. PMID 27275623
- [Background] Jee JH, Ahn HW, Seo KW, Kim SH, Kook YA, Chung KR, Nelson G. En-masse retraction with a preformed nickel-titanium and stainless steel archwire assembly and temporary skeletal anchorage devices without posterior bonding. Korean J Orthod. 2014 Sep;44(5):236-45. doi: 10.4041/kjod.2014.44.5.236. Epub 2014 Sep 25. PMID 25309863
- [Background] Upadhyay M, Yadav S, Nagaraj K, Patil S. Treatment effects of mini-implants for en-masse retraction of anterior teeth in bialveolar dental protrusion patients: a randomized controlled trial. Am J Orthod Dentofacial Orthop. 2008 Jul;134(1):18-29.e1. doi: 10.1016/j.ajodo.2007.03.025. PMID 18617099
- [Background] Kulshrestha RS, Tandon R, Chandra P. Canine retraction: A systematic review of different methods used. J Orthod Sci. 2015 Jan-Mar;4(1):1-8. doi: 10.4103/2278-0203.149608. PMID 25657985
- [Background] Baxmann M, McDonald F, Bourauel C, Jager A. Expectations, acceptance, and preferences regarding microimplant treatment in orthodontic patients: A randomized controlled trial. Am J Orthod Dentofacial Orthop. 2010 Sep;138(3):250.e1-250.e10; discussion 250-1. doi: 10.1016/j.ajodo.2010.03.023. PMID 20816284
- [Background] Lee J, Miyazawa K, Tabuchi M, Sato T, Kawaguchi M, Goto S. Effectiveness of en-masse retraction using midpalatal miniscrews and a modified transpalatal arch: Treatment duration and dentoskeletal changes. Korean J Orthod. 2014 Mar;44(2):88-95. doi: 10.4041/kjod.2014.44.2.88. Epub 2014 Mar 19. PMID 24696825
- [Background] Monga N, Kharbanda OP, Samrit V. Quantitative and qualitative assessment of anchorage loss during en-masse retraction with indirectly loaded miniscrews in patients with bimaxillary protrusion. Am J Orthod Dentofacial Orthop. 2016 Aug;150(2):274-82. doi: 10.1016/j.ajodo.2016.02.014. PMID 27476360
- [Background] Hedayati Z, Shomali M. Maxillary anterior en masse retraction using different antero-posterior position of mini screw: a 3D finite element study. Prog Orthod. 2016 Dec;17(1):31. doi: 10.1186/s40510-016-0143-z. Epub 2016 Oct 3. PMID 27667816
- [Background] Ziegler P, Ingervall B. A clinical study of maxillary canine retraction with a retraction spring and with sliding mechanics. Am J Orthod Dentofacial Orthop. 1989 Feb;95(2):99-106. doi: 10.1016/0889-5406(89)90388-0. PMID 2916474
- [Background] Viecilli RF. Self-corrective T-loop design for differential space closure. Am J Orthod Dentofacial Orthop. 2006 Jan;129(1):48-53. doi: 10.1016/j.ajodo.2004.05.025. PMID 16443478
- [Background] Lee D, Heo G, El-Bialy T, Carey JP, Major PW, Romanyk DL. Initial forces experienced by the anterior and posterior teeth during dental-anchored or skeletal-anchored en masse retraction in vitro. Angle Orthod. 2017 Jul;87(4):549-555. doi: 10.2319/080916-616.1. Epub 2016 Nov 10. PMID 27830931
- [Result] Rhee JN, Chun YS, Row J. A comparison between friction and frictionless mechanics with a new typodont simulation system. Am J Orthod Dentofacial Orthop. 2001 Mar;119(3):292-9. doi: 10.1067/mod.2001.112452. PMID 11244423
- [Derived] Magdi S, Abdelsayed FA, Aboulfotouh MH, Fahim FH. Friction versus frictionless mechanics during maxillary en-masse retraction in adult patients with Class I bimaxillary dentoalveolar protrusion: a randomized clinical trial. Eur J Orthod. 2024 Aug 1;46(4):cjae034. doi: 10.1093/ejo/cjae034. PMID 39011819

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT03261024/Prot_SAP_000.pdf